CLINICAL TRIAL: NCT01174979
Title: Double Blind, Placebo-controlled, Randomized Clinical Trial to Evaluate the Efficacy and Safety of a Transtympanic Treatment of Tinnitus With Caroverine
Brief Title: Caroverin and Inner Ear Diseases
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: due to less patient the study was suspended
Sponsor: Phafag AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-09; 2009-018046-38 (EudraCT Number)
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Tinnitus
Keywords: Morbus Meniere; Sudden hearing loss; Blast injury; Presbyacusis; Chron. Otitis Media
MeSH Terms: conditions — Tinnitus; Hearing Loss, Sudden; Blast Injuries; Presbycusis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caroverin (Experimental)
  Interventions: Drug: Caroverin
- Placebo (Placebo Comparator)
  Interventions: Drug: Caroverin

INTERVENTIONS:
Drug: Caroverin — treatment with eardrops 2 times for 48 hours

SUMMARY:
This trial is a randomized, double blind, placebo controlled study on patients suffering from inner ear diseases with tinnitus as a principal symptom.

The study will investigate the transtympanic treatment with a 1,5 % caroverine solution.

Each patient will undergo treatment for 2 cycles of 48 hours each.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged at least eighteen
* Written consent to take part in the study after receiving information from the trial physician
* One of the following illnesses:

  * Decompensated tinnitus
  * Sudden hearing loss
  * Morbus Menière
  * Blast injury
  * Presbyacusis with Tinnitus
  * Chron. Otitis media

Exclusion Criteria:

* Patients who are not able to give their consent (e.g. dementia, coma, mental disability,…)
* Women of childbearing age who are not using adequate contraception or who are (or plan to become) pregnant (a pregnancy test must be carried out by a doctor once a month in Austria) or are lactating
* If there are solid reasons to doubt that the patient would be willing and able to cooperate
* Known intolerance of/hypersensitivity to caroverine
* Subjects who have taken part in another clinical trial within the 30 days preceding the start of this study or during this study
* Pulse-synchronous tinnitus
* Tinnitus caused by malposition of the jaw bone (bruxism)
* Eardrum perforation
* Subjects who have previously had a barotraumas, diving accidents or decompression sickness
* Retrocochlear hearing disorder
* Patients who have previously had a fracture of the petrous bone
* Subjects suffering from acute or chronic accompanying conditions which severely impede their general health (NYHA stage IV, cancer, HIV etc.)
* Accompanying conditions that according to the current state of scientific knowledge could affect the parameters used in this study to such an extent as to make it impossible to perform an objective assessment of those parameters, particularly ear conditions, including any conditions affecting the other ear or conditions like HI NYHA stage IV, cancer, HIV, Wallenberg Syndrome, massive Hypotension, Glaucoma.)
* Accompanying medication that according to the current state of scientific knowledge are likely to affect the measurement techniques used in this study or the results obtained (cytostatics, aminoglycoside antibiotics, loop diuretics (furosemide, etacrynic acid), psycho pharmaceuticals, muscle relaxants, benzodiazepines, salicylates, quinine, cortisone and/or caroverine within the three days preceding the start of the study)
* Drug treatment for tinnitus or sudden hearing loss (i.v. and oral) within seven days preceding the start of the study where the total duration of the course is less than four weeks
* Diseases or conditions that may be associated with an altered perception or processing of stimuli, e.g. mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
to investigate the efficacy of Caroverin in transtympanic treatment of patients with tinnitus measured by a visual analogue scale. | treatment takes 5 days, follow up examination 4 weeks after

SECONDARY OUTCOMES:
to investigate the time from the start of treatment to an improvement in tinnitus | treatment takes 5 days, follow up examination 4 weeks after
to investigate the efficacy of Caroverin depending the origin of tinnitus | treatment takes 5 days, follow up examination 4 weeks after
to investigate the safety of Caroverin treatment | treatment takes 5 days, follow up examination 4 weeks after
to investigate the impact of Caroverin treatment of quality of life | treatment takes 5 days, follow up examination 4 weeks after

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Elsaesser, Dr., Principal Investigator — Landeskrankenhaus Feldkirch
Locations (1):
- Landeskrankenhaus Feldkirch, Feldkirch, Vorarlberg, Austria